CLINICAL TRIAL: NCT07166965
Title: A Pilot Study of Ketone and Hawthorn Extract Supplementation: Impact on Exercise Capacity, and Heart Function in Patients With Congestive Heart Failure
Brief Title: Ketone and Hawthorn Extract Supplementation in Congestive Heart Failure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: Oncore45335, iRISID-2025-0253
Record Dates: First submitted 2025-07-30; First posted 2025-09-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Congestive Heart Failure(CHF)
Keywords: Heart Failure classified as NYHA Class II or III
MeSH Terms: conditions — Heart Failure | interventions — Ketones

STUDY DESIGN:
Intervention Model Description: Randomization and Intervention At the conclusion of Visit 1, subjects will be randomized to either Group A, B, or C. Group A will be given an over-the-counter Hawthorn extract 500mg capsules to be taken two capsules twice per day. Group B will be given the ketone drink (Ketone-IQ) to take 4 oz (33g) three times per day. Group C will be given 4 oz of a placebo drink and instructed to take it three times per day. All subjects will be instructed to take their intervention for 2 months between the two evaluation visits.
  The randomization and use of supplements will be conducted after all the baseline evaluations are completed: PET MRI, echocardiogram, VO2 MAX.
  The study doctor will decide based on these tests and procedures at this to whether the potential participants would be able to safely participate in the study. The clinical determination of the level of heart disease will be evaluated by the study doctors.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketone supplementation (Experimental): commercially available nutritional ketone monoester
  Interventions: Dietary Supplement: Ketones
- Hawthorn extract (Experimental): commercially available Hawthorn extract
  Interventions: Dietary Supplement: Hawthorn supplement
- Placebo (Placebo Comparator): Placebo supplement
  Interventions: Other: Placebo Control

INTERVENTIONS:
Dietary Supplement: Hawthorn supplement — Hawthorn oral supplement
  Arms: Hawthorn extract
Dietary Supplement: Ketones — ketone oral supplement
  Arms: Ketone supplementation
Other: Placebo Control — Placebo Control, oral supplement
  Arms: Placebo

SUMMARY:
The purpose of this research is to gain a better understanding of whether supplements can improve heart health. There are a number of study procedures and tests that will occur as a part of the research study. There are 3 groups or arms in the study: one group will receive a ketone supplement, one group will receive hawthorn and a third group will receive a placebo that does not contain ketones or hawthorn. The purpose of the study is to learn whether these supplements improve heart heath in patients who have congestive heart failure.

Participants will not know which supplement is received. The study doctor will know. This is called a single blind study. The supplements will provided along with instructions and educational materials. The duration of taking the supplements is approximately 8 weeks and full participation in the study is approximately 3 months. Participants with congestive heart failure will be enrolled through Jefferson Health in Philadelphia, Pennsylvania.

DETAILED DESCRIPTION:
This is a Randomized, placebo-controlled single blind pilot study; the duration of the study enrollment is 24 months. It will be conducted at Thomas Jefferson University, Departments of Integrative Medicine, and Nutritional Sciences; Department of Cardiology. Locations: Marcus Institute Centers of Integrative Health at Villanova and Center City Philadelphia. The enrollment goal is 45: 15 in each study arm, ketone, hawthorn extract, or placebo. The investigators will increase each arm by three for a total of 54 to allow for attrition and early withdrawals. Participants will receive a commercially available Hawthorn extract or nutritional ketone monoester, or placebo.

The Investigators will enroll patients with a diagnosis of stable, ambulatory heart failure, classified by the New York Heart Association (NYHA) as functional Class II or III by their cardiologist and/or by the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or greater than 18 years of age
* Diagnosis of heart failure and be classified as NYHA Class II or III either pre-enrollment or at the time of enrollment: Class II - Patients with cardiac disease resulting in slight limitation of physical activity who are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, or dyspnea (shortness of breath or difficulty breathing).

Class III - Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea (shortness of breath or difficulty breathing).

* Stable guideline directed medical therapy for at least 1 month prior to enrollment, including no changes in maintenance diuretic dosing
* Taking appropriate guideline directed medical therapy as determined by the investigator, who is a heart failure specialist.

Exclusion Criteria

* Patients with Type I DM
* No metal in the body that would prevent undergoing an MRI scan. This includes pacemakers, stents and non-titanium implants that would be contraindicated for an MRI.
* Atrial fibrillation
* Inability to exercise on a treadmill.
* Moderate or greater valvular disease: a condition where the valves of the heart do not function properly.
* Anemia with Hemoglobin <10 g/dL.
* Daily insulin use
* Hypertrophic, infiltrative, or inflammatory cardiomyopathy (a group of heart muscle diseases where the heart muscle becomes abnormally thickened (hypertrophic), invaded by abnormal substances (infiltrative), or inflamed (inflammatory), which can lead to impaired heart function and potential complications like arrhythmias and heart failure.
* Pericardial disease: a general term for conditions that affect the pericardium, the sac that surrounds the heart. Pericardial diseases include pericarditis, pericardial effusion, cardiac tamponade, and constrictive pericarditis..
* Current angina due to clinically significant obstructive epicardial coronary disease. a condition where the major coronary arteries on the surface of the heart (epicardial arteries) become significantly narrowed due to plaque buildup, restricting blood flow to the heart muscle, often causing chest pain and potentially leading to a heart attack.
* Acute coronary syndrome (ACS) refers to a group of conditions where blood flow to the heart is suddenly reduced, causing chest pain or discomfort.
* Coronary intervention within the past 2 months is a medical procedure used to treat ACS by opening a blocked coronary artery, typically done through a minimally invasive technique called percutaneous coronary intervention (PCI).
* Primary pulmonary arteriopathy is also known as pulmonary arterial hypertension (PAH) or primary pulmonary hypertension (PPH), a rare disorder that causes high blood pressure in the pulmonary arteries.
* Known clinically significant lung disease defined as:

  1. Current use of supplemental oxygen, aside from nocturnal O2 for the treatment of obstructive sleep apnea
  2. The use of steroids/antibiotics within the past 6 months for an acute exacerbation of obstructive pulmonary disease
  3. Proximal pulmonary function test (PFT) indicating severe obstructive disease, defined as an FEV1<50% predicted in the context of an FEV1/FVC ratio of <0.70 ("Stage III COPD according to GOLD Criteria: significantly reduced lung function and often accompanied by noticeable symptoms like increased breathlessness, frequent exacerbations, and reduced exercise capacity). (note: only to be used if the subject had PFTs prior to screening)
  4. Proximal 6-minute walk test during which the subject experienced desaturation (<94%) without subsequent normal study.
* Ischemia on stress testing without subsequent revascularization or left heart catheterization showing non-obstructive epicardial coronary disease.
* Significant liver diseases impact on synthetic function or volume control.
* Uncontrolled hypertension: BP >180/110 at baseline.
* Estimated glomerular filtration rate (eGFR) eGFR <30 mL/min/173m2 indicating reduced kidney function
* Creatinine level of Cr >2.5 (2.5 mg/dL) is an indicator of stage 2 chronic kidney disease (CKD).
* Current Alcohol dependence
* Current substance use disorder.
* Chronic narcotic use that cannot be interrupted
* Pregnant or lactating females
* Subject has a medical, mental or psychiatric disorder or physical condition that could reasonably be expected to interfere with the assessment of cardiac symptoms, or with any of the study assessments or study procedures including the PET-MRI imaging, VO2 Max, Echocardiogram ultrasound, blood samples that would put the study participant at great risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Measure and Compare Changes in Myocardial Function: exercise capacity | From baseline enrollment evaluations with functional measures to the end of supplementation at 8 weeks and evaluations afterwards at weeks 10 to 12.
  Compare outcomes of functional measures - exercise capacity as measured by oxygen consumption at peak and anaerobic threshold (VO2peak and VO2at) and exercise duration.
  Exercise capacity is measured objectively through laboratory Cardiopulmonary Exercise Tests (CPETs) combined metrics which use equipment to monitor heart rate, breathing, and oxygen consumption; with VO2 peak setting the ceiling for endurance and VO2AT.
  Exercise capacity, measured by oxygen consumption (VO2), to measure the body's ability to take in and use oxygen during exercise, with VO2 peak representing the maximum capacity reached and VO2 at the anaerobic threshold (VO2AT) at rest and during peak exercise following approximately 2 months of receiving the respective supplementation or placebo.
Measure and Compare Changes in Myocardial Function: Structure and heart function | From baseline enrollment evaluations with functional measures to the end of supplementation at 8 weeks and evaluations afterwards at weeks 10 to 12.
  Compare outcomes of functional measures as measured by changes in myocardial function (evaluate the structure and function of the heart and blood vessels) at rest as measured by Cardiac Magnetic Resonance Imaging (cMRI) indexes of Left ventricular ejection fraction (LVEF) and Right Ventricular Ejection Fraction (RVEF) and myocardial performance at peak exercise (cardiac output [CO] and LVEF) as measured by echocardiogram at rest and during peak exercise following approximately 2 months of receiving the respective supplementation or placebo.

SECONDARY OUTCOMES:
Measure and Compare Changes Associated with Supplementation using FDG PET and Cardiac MRI | From baseline enrollment evaluations with functional measures to the end of supplementation at 8 weeks and evaluations afterwards at weeks 10 to 12.
  Compare changes associated with the respective nutraceutical supplementation in cardiac glucose uptake as measured by Fluoro deoxy glucose Positron Emission Tomography (FDG PET) and cardiac function as measured by cardiac MRI.
Measure and Compare Changes Associated with Cardiac Metabolism using FDG PET and Cardiac MRI | From baseline enrollment evaluations with functional measures to the end of supplementation at 8 weeks and evaluations afterwards at weeks 10 to 12.
  Compare changes associated with the respective nutraceutical supplementation in cardiac glucose uptake as measured by Fluoro deoxy glucose Positron Emission Tomography (FDG PET) and cardiac function as measured by cardiac MRI.

OTHER OUTCOMES:
Height in inches | From baseline enrollment evaluations with functional measures
  Height will be collected at baseline (not expected to change).
Weight in pounds | From baseline enrollment evaluations with functional measures to the end of supplementation at 8 weeks and evaluations afterwards at weeks 10 to 12.
  Weight will be collected at baseline and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Newberg, MD, Principal Investigator — Thomas Jefferson University, Marcus Institute
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No